CLINICAL TRIAL: NCT03667105
Title: Evaluation of Two Types of Matrix (Mucograft® and Mucoderm®) Associated With Coronally Advanced Flap for the Treatment of Single Gingival Recessions: Randomized Clinical Trial
Brief Title: Evaluation of Two Types of Matrix (Mucograft® and Mucoderm®) Associated With Coronally Advanced Flap
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Estadual Paulista Júlio de Mesquita Filho (Other)
Responsible Party: Principal Investigator, Mauro Pedrine Santamaria, Assistant Professor, Universidade Estadual Paulista Júlio de Mesquita Filho
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MC - XDM
Record Dates: First submitted 2018-09-10; First posted 2018-09-12 (Actual); Last update posted 2020-05-01 (Actual); Status verified 2020-04

CONDITIONS: Gingival Recession
MeSH Terms: conditions — Gingival Recession | interventions — Mucograft; Mucoderm

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CAF+XDM (Experimental): CAF treatment will be performed by starting with two divergent releasing incisions lateral to the recessed area. A sulcular incision will be made to unite the releasing incisions and the flap will be raised beyond the mucogingival junction (MGJ) in split-full-split thickness. Additionally, this group will receive the xenogenous dermal collagen matrix graft (AXDM - Mucoderm®, Botiss,) on the recessed area before the sutures. Then, the flap will be coronally positioned and sutured to completely cover the graft.
  Interventions: Procedure: CAF; Other: XDM
- CAF+MC (Experimental): CAF treatment will be performed by starting with two divergent releasing incisions lateral to the recessed area. A sulcular incision will be made to unite the releasing incisions and the flap will be raised beyond the mucogingival junction (MGJ) in split-full-split thickness. Additionally, this group will receive the xenogenous collagen matrix graft (Mucograft®, Geistlich Pharma) on the recessed area before the sutures. Then, the flap will be coronally positioned and sutured to completely cover the graft.
  Interventions: Procedure: CAF; Other: MC
- CAF (Active Comparator): CAF treatment will be performed by starting with two divergent releasing incisions lateral to the recessed area. A sulcular incision will be made to unite the releasing incisions and the flap will be raised beyond the mucogingival junction (MGJ) in split-full-split thickness. Then, the flap will be coronally positioned and sutured to completely cover the graft. This group will be the control group.
  Interventions: Procedure: CAF

INTERVENTIONS:
Procedure: CAF — Periodontal surgical technique to treat gingival recessions.
  Other Names: Periodontal plastic surgery
Other: MC — Xenogenous graft placed in the surgical site.
  Other Names: Xenogenous collagen matrix graft (Mucograft®)
  Arms: CAF+MC
Other: XDM — Xenogenous dermal collagen graft placed in the surgical site.
  Other Names: Xenogenous dermal collagen matrix graft (Mucoderm®)
  Arms: CAF+XDM

SUMMARY:
The aim of this study is to evaluate clinically the results of two types of matrix (Geistlich Mucograft® and Mucoderm®) associated with CAF technique for the treatment of gingival recessions.

DETAILED DESCRIPTION:
This is a prospective, parallel and controlled clinical trial. The population that will be evaluated in the study will be selected at Institute of Science and Technology (ICT), São José dos Campos, College of Dentistry.

Seventy-five patients presenting gingival recession will be divided in 3 groups:

* Group CAF + XDM (25): Periodontal surgery for root coverage through coronally advanced flap technique plus xenogenous dermal matrix graft Mucoderm®.
* Group CAF + MC (25): Periodontal surgery for root coverage through coronally advanced flap technique plus xenogenous collagen matrix graft Mucograft®.
* Group CAF (25): Periodontal surgery for root coverage through coronally advanced flap alone.

All surgeries will be performed by a single operator (MPS) at the dental clinic of ICT. Two horizontal incisions will be made at right angles to the adjacent interdental papillae, without interfering with gingival margins of neighboring teeth. Two oblique vertical incisions will be extended beyond the mucogingival junction and a trapezoidal mucoperiosteal flap will be raised up to the mucogingival junction. After, a split-thickness flap will be extended apically, releasing the tension and favoring coronal positioning of the flap. The exposed root surface will be scaled and planed. After the root planning procedures are performed, the epithelial layer from incised papillae will be removed to expose the connective tissue. After this, the group in which the participant is inserted will be revealed to the surgeon. The grafts will be used according to the producers' instructions. In the CAF + MD group, the matrix will be placed without previous hydration with saline solution, whereas in the CAF + XDM group the matrix will be hydrated with sterile saline for 10 minutes. In both grafts groups, the matrix will be cut into the desired dimensions to cover the entire surface of the root and around the bone, being positioned at the CEJ level. The matrix will be sutured independently of the flap, with the porous surface in contact with the tooth and bone, while the smooth surface will be facing the flap. Then, the flap will be coronally positioned and sutured to completely cover the graft. After the surgical procedure, the patients will receive the appropriate postoperative recommendations and sutures will be removed after 10 to 14 days of the surgical procedure.

Clinical parameters will be assessed at baseline and 3 and 6 months postoperatively.

Quantitative data were recorded as mean ± standard deviation (SD), and normality was tested using Shapiro-Wilk tests. The probing depth (PD), relative gingival recession (RGR), clinical attachment level (CAL), keratinized tissue thickness (KTT), keratinized tissue width (KTW), aesthetic (A), postoperative discomfort (PD), dentin hypersensitivity (DH) and tissue edema (TE) values will be examined variance test. Patients' esthetics and discomfort measures using a visual analog scale (VAS) will be analyzed by T-tests. The frequency of complete root coverage will be compared using χ2 tests. Intergroup root coverage esthetic score (RES) comparisons will be performed with a T-test.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting Miller class I or II gingival recession in the maxillary canines or premolars;
* Teeth included in the study should present pulp vitality and no associated with carious or cervical lesion;
* Patients presenting no signs of active periodontal disease and full-mouth plaque and bleeding score ≤ 20%;
* Probing depth ˂ 3 mm in the included and adjacent teeth, presenting no signs of bleeding or attachment loss;
* Patients older than 18 years old;
* Patients who agreed to participate and signed an informed consent form.

Exclusion Criteria:

* Patients with systemic problems (cardiovascular, blood dyscrasias, immunodeficiency, and diabetes, among others) that will contraindicate the surgical procedure;
* Patients taking medications known to interfere with the wound healing process or that contraindicate the surgical procedure;
* pregnant or lactating women;
* Smokers;
* Patients who underwent periodontal surgery in the area of interest;
* Patients with orthodontic therapy in progress.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2018-08-15 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2020-02-25 (Actual)

PRIMARY OUTCOMES:
Percentage of defect coverage | 6 months
  Percentage mean (%) of root surface covered by the surgical treatment, measured through a periodontal probe.

SECONDARY OUTCOMES:
Root coverage esthetic score | 6 months
  This analysis will be performed through the Root Coverage Aesthetics Scale (RES, cairo et al., 2009), by 3 blinded and independent examiners at the 6-month post-operative assessment. The RES method uses a "score" that evaluates the following parameters:
  * Level of the gingival margin (0=failure of the root covering, 3=partial covering, 6=total covering);
  * Marginal tissue contour (0=irregular contour, 1=normal contour);
  * Soft tissue texture (0=presence of scar or keloid; 1=absence of scar or keloid);
  * Mucogingival junction alignment: (0=mucogingival line not aligned with the line of the neighboring teeth; 1=mucogingival line aligned with the line of the neighboring teeth);
  * Gingival color (0=color of gingival tissue different from the neighboring tissues; 1=color of treated gingival tissue equal to neighboring tissues).
  According to the sum of scores received, the teeth will be considered: aesthetic (score=10), partially aesthetic (score= 1-9) or without aesthetic (score=0).
Evaluation of root dentine hypersensitivity with the air blow test | 6 months
  The assessment of root sensitivity will be performed by applying a blow of air in the region of the surgical procedure for 5 seconds. The patient should mark on a Visual Analogue Scale (VAS) the perceived sensitivity. On this visual scale (range 0-10), the extreme "0" represents "none discomfort or sensitivity" and the extreme "10" represents "extreme discomfort or sensitivity". Thus, higher values represent a worse outcome.
Evaluation of patient recovery through the report of discomfort and postoperative pain | 7 days
  At the end of the first post-operative week (7 days) the patients will receive a questionnaire with questions about the occurrence of discomfort and postoperative pain, that will be evaluated by means of a Visual Analog Scale (VAS). On this visual scale (range 0-10), the extreme "0" represents "none discomfort or pain" and the extreme "10" represents "extreme discomfort or pain". Thus, higher values represent a worse outcome. In addition, patients were asked to report the number of analgesics tablets ingested during that week.
Aesthetic evaluation according to patient through Visual Analog Scale (EVA) | 6 months
  Aesthetic evaluation according to the opinion of the patient will be performed in the baseline and at the 6-month post-operative assessment. Looking at a mirror, the patient will visualize the area of gingival surgery and mark in a Visual Analogue Scale (EVA) the aesthetic of the element in question. On this visual scale, the left extreme represents "very ugly" and the right extreme represents "very beautiful". Thus, closer values of "very beautiful" will represent better outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Mauro P Santamaria, PhD, Principal Investigator — ICT-UNESP
Locations (1):
- Laís Fernanda Ferreira Ferraz, São José dos Campos, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Moreira ARO, Santamaria MP, Silverio KG, Casati MZ, Nociti Junior FH, Sculean A, Sallum EA. Coronally advanced flap with or without porcine collagen matrix for root coverage: a randomized clinical trial. Clin Oral Investig. 2016 Dec;20(9):2539-2549. doi: 10.1007/s00784-016-1757-8. Epub 2016 Feb 26. PMID 26917493
- [Background] Tonetti MS, Cortellini P, Pellegrini G, Nieri M, Bonaccini D, Allegri M, Bouchard P, Cairo F, Conforti G, Fourmousis I, Graziani F, Guerrero A, Halben J, Malet J, Rasperini G, Topoll H, Wachtel H, Wallkamm B, Zabalegui I, Zuhr O. Xenogenic collagen matrix or autologous connective tissue graft as adjunct to coronally advanced flaps for coverage of multiple adjacent gingival recession: Randomized trial assessing non-inferiority in root coverage and superiority in oral health-related quality of life. J Clin Periodontol. 2018 Jan;45(1):78-88. doi: 10.1111/jcpe.12834. Epub 2017 Nov 21. PMID 29087001
- [Background] Cardaropoli D, Tamagnone L, Roffredo A, Gaveglio L. Treatment of gingival recession defects using coronally advanced flap with a porcine collagen matrix compared to coronally advanced flap with connective tissue graft: a randomized controlled clinical trial. J Periodontol. 2012 Mar;83(3):321-8. doi: 10.1902/jop.2011.110215. Epub 2011 Jul 1. PMID 21721988
- [Background] Sangiorgio JPM, Neves FLDS, Rocha Dos Santos M, Franca-Grohmann IL, Casarin RCV, Casati MZ, Santamaria MP, Sallum EA. Xenogenous Collagen Matrix and/or Enamel Matrix Derivative for Treatment of Localized Gingival Recessions: A Randomized Clinical Trial. Part I: Clinical Outcomes. J Periodontol. 2017 Dec;88(12):1309-1318. doi: 10.1902/jop.2017.170126. Epub 2017 Jul 28. PMID 28753100